CLINICAL TRIAL: NCT04387500
Title: Single-arm Phase II Clinical Trial to Evaluate the Initial Efficacy and Safety of Sintilimab Injection Combined With Inlyta in Fumarate Hydratase- Deficient Renal Cell Carcinoma
Brief Title: Sintilimab Injection Combined With Inlyta in Fumarate Hydratase- Deficient Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor of Department of Urology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190813
Record Dates: First submitted 2019-08-15; First posted 2020-05-14 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Renal Cell; Fumarate Hydratase Deficiency; Immunotherapy
Keywords: Sintilimab; Inlyta
MeSH Terms: conditions — Carcinoma, Renal Cell; Fumaric aciduria | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab injection combined with Inlyta (Experimental): Sintilimab injection 10ml: 100mg, 200mg intravenously, once every three weeks. Course of treatment: discontinue medication when the disease progresses clinically or radiologically.
  Inlyta 5mg orally, twice a day. Course of treatment: continue treatment as long as a clinical benefit is observed, or until an unacceptable toxicity is present that cannot be controlled by combination or dose adjustment.
  In the whole research process, if the disease progresses, the attending doctor has the right to carefully choose other anti-tumor methods, including radiotherapy, chemotherapy and other targeted drugs.
  Interventions: Drug: Sintilimab injection plus Inlyta treatment

INTERVENTIONS:
Drug: Sintilimab injection plus Inlyta treatment — Combined Sintilimab injection and Inlyta treatment in FH-deficient RCC

SUMMARY:
This is a single-arm phase II clinical trial to evaluate the initial efficacy and safety of Sintilimab injection combined with Inlyta in fumarate hydratase-deficient renal cell carcinoma.

DETAILED DESCRIPTION:
Our previous genetic research as well as other published data indicated the possible well response to combination of immunotherapy with targeted therapy in FH-deficient renal cell carcinoma, therefore the investigators intented to perform this single-arm phase II clinical trial to evaluate the initial efficacy and safety of Sintilimab injection combined with Inlyta in FH-deficient renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, no gender limitation;
2. Histopathological confirmed RCC, and diagnosed as FH-dRCC by Sanger or NGS sequencing after being included in preliminary IHC screening;
3. The patients incuded must be diagnosed with metastatic RCC or TNM stage IV (according to the 2009 TNM staging system), with distant metastasis confirmed by radiology or pathology.
4. Have not received systemic treatment, including cytokines, targeted drugs, or other experimental drugs, or have received targeted drugs (within the range of 1st-line targeted drugs recommended by NCCN2022 for renal cancer) with single drug treatment for less than 1 month and have completed the washout period. ECOG score ≤ 2;
5. Life expectancy ≥ 3 months;
6. Signed written informed consent form and willing and able to comply with scheduled visits and other requirements of the study；
7. Agree to collect tumor tissue and blood samples required for this study and apply the samples to relevant studies;
8. Adequate organ and bone marrow function: absolute neutrophil count (ANC): ≥1×109/L, platelet count (PLT) ≥50×109/L, hemoglobin content (HGB) ≥80g/L; Liver function: total bilirubin (TBIL) ≤3×normal upper limit (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤5×ULN, albumin ≥20g/L; Renal function: serum creatinine (Cr) ≤3×ULN.

Exclusion Criteria:

1. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA4 antibody, or any other antibodies or drugs specifically targeting co-stimulatory or checkpoint pathways of T cells;
2. Active brain metastasis;
3. Other malignancy with primary site or histological type different from tumors evaluated in this study within 2 years of personal history, except skin basal cell carcinoma, squamous cell carcinoma or adequately treated cervical carcinoma in situ;
4. Underwent major operation (craniotomy, thoracotomy or laparotomy) within 4 weeks of the first dose of study medication or with severe trauma;
5. Received systemic treatment with corticosteroids (> 10mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks of first dose. Inhaled or topical steroids and adrenal replacement steroid doses are permitted in the absence of active autoimmune disease.
6. Known or suspected active autoimmune disease (congenital or acquired), including interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroiditis, etc. Patients with type I diabetes, hypothyroidism that only requires systemic treatment (including vitiligo, psoriasis, alopecia, etc.), or conditions that are not expected to recur in the absence of external triggers are eligible to participate in this study; Known history of allogeneic organ (except corneal transplantation) or allogeneic hemopoietic stem cell transplantation;
7. Known allergy or hypersensitivity to any monoclonal antibodies or any components used in their preparation;
8. Uncontrolled concomitant disease, including but not limited to:

   1. Active or poorly controlled severe infection;
   2. Human Immunodeficiency Virus (HIV) infection (HIV antibody positive);
   3. Known acute or chronic active hepatitis B infection (HBsAg positive and HBV DNA>1*103/ml), or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA>15IU/ml);
   4. Active tuberculosis;
9. Symptomatic congestive heart failure (New York Heart Association grade III-IV) or symptomatic, poorly controlled arrhythmia;
10. Poorly controlled arterial hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg) with standard treatment;
11. Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke and transient ischemic attack, within 6 months of enrollment;
12. Diseases that require anticoagulant treatment with warfarin (coumarin);
13. Poorly controlled hypercalcemia (Ca2+ > 1.5mmol/L, or serum calcium > 12mg/dL, or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring bisphosphate treatment;
14. Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study;
15. Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  objective response rate
PFS | 3 years
  progression-free survival

SECONDARY OUTCOMES:
OS | 3 years
  overall survival
EQ-5D-5L | Up to 36 months
  EQ-5D-5L score change over time from baseline to disease progression. The EQ-5D-5L is consisted of five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Higher scores indicate poorer health.
FKSI-19 | Up to 36 months
  FKSI-19 score change over time from baseline to disease progression. The scale of FKSI-19 is from 0 to 48, and higher scores indicate worse quality of life.
DCR | 3 years
  Disease control rate
Duration of response | 3 years
  time from the first occurrence of treatment response (CR or PR) to disease progression or death
VAS | 3 years
  VAS pain score change over time from baseline to disease progression. The scale of VAS is from 0-10, and higher scores indicate worse symptom of pain.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data would be available starting from the time when summary data are published or otherwise made available, for 3 years.
Access Criteria: Other researchers access the data by sending an email to our PI.

REFERENCES:
- [Background] Tomlinson IP, Alam NA, Rowan AJ, Barclay E, Jaeger EE, Kelsell D, Leigh I, Gorman P, Lamlum H, Rahman S, Roylance RR, Olpin S, Bevan S, Barker K, Hearle N, Houlston RS, Kiuru M, Lehtonen R, Karhu A, Vilkki S, Laiho P, Eklund C, Vierimaa O, Aittomaki K, Hietala M, Sistonen P, Paetau A, Salovaara R, Herva R, Launonen V, Aaltonen LA; Multiple Leiomyoma Consortium. Germline mutations in FH predispose to dominantly inherited uterine fibroids, skin leiomyomata and papillary renal cell cancer. Nat Genet. 2002 Apr;30(4):406-10. doi: 10.1038/ng849. Epub 2002 Feb 25. PMID 11865300
- [Background] Isaacs JS, Jung YJ, Mole DR, Lee S, Torres-Cabala C, Chung YL, Merino M, Trepel J, Zbar B, Toro J, Ratcliffe PJ, Linehan WM, Neckers L. HIF overexpression correlates with biallelic loss of fumarate hydratase in renal cancer: novel role of fumarate in regulation of HIF stability. Cancer Cell. 2005 Aug;8(2):143-53. doi: 10.1016/j.ccr.2005.06.017. PMID 16098467
- [Background] Mullen AR, Wheaton WW, Jin ES, Chen PH, Sullivan LB, Cheng T, Yang Y, Linehan WM, Chandel NS, DeBerardinis RJ. Reductive carboxylation supports growth in tumour cells with defective mitochondria. Nature. 2011 Nov 20;481(7381):385-8. doi: 10.1038/nature10642. PMID 22101431
- [Background] Ooi A, Wong JC, Petillo D, Roossien D, Perrier-Trudova V, Whitten D, Min BW, Tan MH, Zhang Z, Yang XJ, Zhou M, Gardie B, Molinie V, Richard S, Tan PH, Teh BT, Furge KA. An antioxidant response phenotype shared between hereditary and sporadic type 2 papillary renal cell carcinoma. Cancer Cell. 2011 Oct 18;20(4):511-23. doi: 10.1016/j.ccr.2011.08.024. PMID 22014576
- [Background] Voss MH, Molina AM, Chen YB, Woo KM, Chaim JL, Coskey DT, Redzematovic A, Wang P, Lee W, Selcuklu SD, Lee CH, Berger MF, Tickoo SK, Reuter VE, Patil S, Hsieh JJ, Motzer RJ, Feldman DR. Phase II Trial and Correlative Genomic Analysis of Everolimus Plus Bevacizumab in Advanced Non-Clear Cell Renal Cell Carcinoma. J Clin Oncol. 2016 Nov 10;34(32):3846-3853. doi: 10.1200/JCO.2016.67.9084. PMID 27601542
- [Background] Kusmartsev S, Eruslanov E, Kubler H, Tseng T, Sakai Y, Su Z, Kaliberov S, Heiser A, Rosser C, Dahm P, Siemann D, Vieweg J. Oxidative stress regulates expression of VEGFR1 in myeloid cells: link to tumor-induced immune suppression in renal cell carcinoma. J Immunol. 2008 Jul 1;181(1):346-53. doi: 10.4049/jimmunol.181.1.346. PMID 18566400
- [Background] Wallin JJ, Bendell JC, Funke R, Sznol M, Korski K, Jones S, Hernandez G, Mier J, He X, Hodi FS, Denker M, Leveque V, Canamero M, Babitski G, Koeppen H, Ziai J, Sharma N, Gaire F, Chen DS, Waterkamp D, Hegde PS, McDermott DF. Atezolizumab in combination with bevacizumab enhances antigen-specific T-cell migration in metastatic renal cell carcinoma. Nat Commun. 2016 Aug 30;7:12624. doi: 10.1038/ncomms12624. PMID 27571927
- [Background] Najjar YG, Rayman P, Jia X, Pavicic PG Jr, Rini BI, Tannenbaum C, Ko J, Haywood S, Cohen P, Hamilton T, Diaz-Montero CM, Finke J. Myeloid-Derived Suppressor Cell Subset Accumulation in Renal Cell Carcinoma Parenchyma Is Associated with Intratumoral Expression of IL1beta, IL8, CXCL5, and Mip-1alpha. Clin Cancer Res. 2017 May 1;23(9):2346-2355. doi: 10.1158/1078-0432.CCR-15-1823. Epub 2016 Oct 31. PMID 27799249
- [Result] Zhang X, Liu H, Zhang Y, et al. Phase II, multi-center study of sintilimab in combination with axitinib in patient with advanced fumarate hydratase-deficient renal cell carcinoma. Presented at: 2023 AUA Annual Meeting; April 28-May 1, 2023; Chicago, IL. Abstract PD24-09.
- [Derived] Zhang X, Liu H, Liang J, Zhao J, Wang Y, Chen Y, Kang D, Chen Q, Zhang Y, Yin X, Zeng Y, Wang Z, Sheng X, Yao X, Gong K, Liu X, Chen Z, Qiu M, Chen W, Wang Z, Luo G, Zhou T, Yang N, Pan X, Nie L, Zhang M, Chen J, Zhao J, Hu X, Xu L, Tang B, Dai J, Liu H, Ni Y, Huang R, Wei Q, Li X, He Q, Liu J, Shen P, Chen N, Liu Z, Sun G, Yao J, Zeng H. Sintilimab Plus Axitinib for Advanced Fumarate Hydratase-Deficient Renal Cell Carcinoma: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2025 Oct 1;11(10):1169-1177. doi: 10.1001/jamaoncol.2025.2497. PMID 40810951

DOCUMENTS (1):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04387500/Prot_000.pdf